CLINICAL TRIAL: NCT03553173
Title: A Randomized Open-label Parallel-group Trial is to Analyze the Efficacy and the Efficiency of the Social-Local-Mobile (So-Lo-Mo) Intervention Applied to the Smoking Cessation Process.
Brief Title: So-Lo-Mo Intervention Applied to the Smoking Cessation Process
Acronym: So-Lo-Mo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: European Commission (Other); Andaluz Health Service (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFB-APP_EC-2016-01
Record Dates: First submitted 2018-05-02; First posted 2018-06-12 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Smoking Cessation; Health Behavior; Lifestyle-related Condition
Keywords: Smoking Cessation; App; Decision Support System
MeSH Terms: conditions — Smoking Cessation; Health Behavior; Mental Disorders; Alzheimer Disease | interventions — Bupropion; Varenicline

STUDY DESIGN:
Intervention Model Description: A randomized open-label parallel-group trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Subjects undergoing usual psycho-pharmacological treatment for smoking cessation.
  Prescribed treatments:
  * Bupropion pills + Psychological advice
  * Varenicline pills + Psychological advice
  Interventions: Behavioral: Psychological advice; Drug: Bupropion Pill; Drug: Varenicline Pill
- Intervention (Experimental): Subjects undergoing usual psycho-pharmacological treatment for smoking cessation plus a smart phone App.
  Prescribed treatments:
  * Bupropion pills + Psychological advice + So-Lo-Mo
  * Varenicline pills + Psychological advice + So-Lo-Mo
  Interventions: Other: So-Lo-Mo; Behavioral: Psychological advice; Drug: Bupropion Pill; Drug: Varenicline Pill

INTERVENTIONS:
Other: So-Lo-Mo — So-Lo-Mo is an innovative intervention based on mobile technologies and its capacity to trigger behavioral changes. In this sense, the App is a complement to pharmacological therapies to quit smoking providing personalised motivational messages, physical activity monitoring, lifestyle advices and distractions (mini-games) to help pass the cravings. The main objective of this App is to improve patient's adherence to the smoking cessation process making use of behavioral techniques in the form of motivational messages and/or Short Message Service (SMS).
  Other Names: SoLoMo
  Arms: Intervention
Behavioral: Psychological advice — Provision of information about smoking and smoking cessation process, as well as supporting behavioral changes through the provision of new skills and strategies. The most used methods are the motivational interview and the cognitive-behavioral therapy
  Other Names: Behavioral
Drug: Bupropion Pill — Formulated as a 150 mg long discharge pill, usually being prescribed a daily dose of 300 mg, except for week one which would be prescribed 150 mg per day. The usual length of the treatment ranges from 7 to 9 weeks. However, 12 weeks treatments could be prescribed for severe cases of smokers.
  Other Names: Bupropion
Drug: Varenicline Pill — Formulated as 0,5 mg and 1 mg pills, and the dose should be progressively incremented during the first days in order to facilitate tolerance. The recommended length of the treatment is 12 weeks, although longer treatments could be necessary for severe smokers.
  Other Names: Varenicline

SUMMARY:
This is a randomized open-label parallel-group trial. 240 subjects will be recruited during 8 months and a 12 months follow-up will be carried out for each one of them. The sample will split in two groups: control group (n=120) who will receive usual psycho-pharmacological therapy and the intervention group (n=120) who will receive usual therapy plus So-Lo-Mo app.

DETAILED DESCRIPTION:
The main objective of this study is to analyze the efficacy and efficiency of the So-Lo-Mo intervention applied to the smoking cessation process compared to usual care.

Secondary objectives are:

1. To monitor usual psycho-pharmacological therapies (bupropion, varenicline and behavioural therapy).
2. To monitor healthy lifestyle and physical exercise habits.

ELIGIBILITY:
Inclusion Criteria:

* Smoking population attending to the Smoking Cessation Unit of "Virgen del Rocío" University Hospital.
* Subjects >18 years old who want to give up smoking.
* Android-based smart phone availability.
* Ability to interact with the smart phone.
* To sign an Informed Consent Form.

Exclusion Criteria:

* Subjects had some previous adverse effects related to the pharmacological treatment included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Efficacy: Smoking abstinence rate | 1 year
  Smoking abstinence rate at 1 year measured by means of exhaled Carbon Monoxide (CO) and urinary cotinine tests. Subjects with cotinine concentrations >200 ng/ml or CO >6 ppm will be considered as smokers.
Efficiency: Incremental Cost-Effectiveness Ratio | 1 year
  Expressed in terms of Incremental Cost-Effectiveness Ratio (ICER), calculated by dividing the difference in total costs between the intervention group and the control group by the difference in Quality-Adjusted Life Year (QALY) between both groups. Costs associated to control and intervention groups will include healthcare resources utilization measured in terms of specialist consultations related to the smoking cessation process. Costs of pharmacological treatment and time employed by healthcare professionals during the design phase will also be taken into account. Benefit for patients will be expressed in terms of QALY. EuroQol-5D-5L questionnaire will be used to estimate QALY.

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events [Safety] | 1 year
  To monitor usual pharmacological therapies (bupropion and varenicline) in order to gather the incidence of related adverse events reported. Safety will be measured as the number of adverse events related to pharmacological therapies. The following adverse events have been identified related to each pharmacological therapy:
  Varenicline: Nausea, vomit, headache, insomnia, abnormal dreams, constipation and flatulence.
  Bupropion: insomnia, headache, dryness in the mouth, alteration of taste, skin reactions, convulsions, cardiovascular side effects and severe skin reactions.
International Physical Activity Questionnaire (IPAQ27) score [Physical activity] | From baseline (first evaluation in the study) to 1 year after
  Physical activity will be measured in terms of the International Physical Activity Questionnaire (IPAQ27) score calculation at baseline (first evaluation in the study) and at the end of the intervention (after 1 year of follow-up). The result is expressed as metabolic equivalent (MET)-minutes per week. Interpretation:
  * Low: Individuals who not meet criteria for categories 2 or 3 are considered 'low'
  * Moderate: 3 or more days of vigorous-intensity activity of at least 20 minutes per day OR 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day OR 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum Total physical activity of at least 600 MET-minutes/week
  * High: vigorous-intensity activity on at least 3 days achieving a minimum Total physical activity of at least 1500 MET-minutes/week
Body Mass Index (BMI) in kg/m^2 [Healthy lifestyle] | From baseline (first evaluation in the study) to 1 year after
  Healthy lifestyle will be measured in terms of the subject's BMI (weight in kg / height in m^2) at baseline (first evaluation in the study) and at the end of the intervention (after 1 year of follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Ortega-Ruiz, MD, PhD, Principal Investigator — Virgen del Rocío University Hiospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Carrasco-Hernandez L, Jodar-Sanchez F, Nunez-Benjumea F, Moreno Conde J, Mesa Gonzalez M, Civit-Balcells A, Hors-Fraile S, Parra-Calderon CL, Bamidis PD, Ortega-Ruiz F. A Mobile Health Solution Complementing Psychopharmacology-Supported Smoking Cessation: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Apr 27;8(4):e17530. doi: 10.2196/17530. PMID 32338624
- [Derived] Jodar-Sanchez F, Carrasco Hernandez L, Nunez-Benjumea FJ, Mesa Gonzalez MA, Moreno Conde J, Parra Calderon CL, Fernandez-Luque L, Hors-Fraile S, Civit A, Bamidis P, Ortega-Ruiz F. Using the Social-Local-Mobile App for Smoking Cessation in the SmokeFreeBrain Project: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Dec 6;7(12):e12464. doi: 10.2196/12464. PMID 30522992

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03553173/Prot_SAP_000.pdf